CLINICAL TRIAL: NCT07083596
Title: The Efficacy of Fermented Milk Drink With Lacticaseibacillus Paracasei Strain Shirota (LcS) on Relieving Constipation-Related Symptoms of Filipino Adults
Brief Title: Efficacy of LcS-Fermented Milk on Constipation-Related Symptoms in Filipino Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santo Tomas (Other)
Collaborators: Yakult Honsha Co., LTD (Industry)
Responsible Party: Principal Investigator, Diane S. Mendoza-Sarmiento, Principal Investigator, University of Santo Tomas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-2025-06-084-CT-AP; 2025-06-084-CT-R1 (Other: University of Santo Tomas REC)
Record Dates: First submitted 2025-07-06; First posted 2025-07-24 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Constipation; Gastrointestinal Discomfort
Keywords: probiotic; Lacticaseibacillus paracasei strain Shirota; constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Data encoder, Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Probiotic drink with Lacticaseibacillus paracasei strain Shirota will be consumed once per day for four weeks
  Interventions: Other: Experimental: Probiotic with LcS
- Control (Placebo Comparator): Brochure containing recommendations to improve constipation will be provided at the end of study.
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental: Probiotic with LcS — Probiotic drink with LcS will be consumed once per day for four weeks
  Arms: Probiotic
Other: Control — Brochure containing recommendations to improve constipation will be provided at end of study.
  Arms: Control

SUMMARY:
The primary purpose of this study is to investigate whether the consumption of a probiotic drink (with Lacticaseibacillus paracasei strain Shirota (LcS)) relieves constipation-related symptoms of Filipino adults, specifically its effect on stool consistency, frequency, and duration, and on gastrointestinal discomfort.

DETAILED DESCRIPTION:
The goal of this clinical trial is to test if probiotic drink with LcS consumption can improve constipation-related symptoms. The main question[s] it aims to answer are:

* Will a probiotic drink with LcS improve stool consistency after four weeks?
* Will a probiotic drink with LcS improve stool frequency and duration after four weeks?
* Will a probiotic drink with LcS improve gastrointestinal discomfort after four weeks?

Participants will consume probiotic drink with LcS once a day for four weeks while maintaining their usual physical activity. Researchers will compare the control group and the probiotic group to see if there are differences in stool consistency, frequency and duration, and gastrointestinal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Filipino adult male or female aged 18 to 59 years old
* Apparently healthy adults with constipation-related symptoms of hard to lumpy stools (Bristol Stool Form Scale 1-2) in 25% or more of defecations in a week
* With cold storage at home

Exclusion Criteria:

1. Habitual intake of food items containing probiotics and prebiotics as food supplements (previous 3 months, at least three times per week)
2. Constipation due to organic or neurologic origin
3. High fiber intake (>30 g/day)
4. Pregnant or lactating
5. Allergy to dairy products and/or lactose intolerance
6. Use of laxatives, anticholinergics and medications for constipation or diarrhea within the past three months
7. Use of antibiotics within the past two weeks
8. Presence of chronic diseases such as diabetes mellitus and its complications, cardiovascular diseases, kidney problems
9. GI condition that may interfere with the evaluation of the outcome such as hemorrhoids, intestinal obstruction and inflammatory bowel diseases
10. Recent history of any gastrointestinal surgery
11. Have pre-existing medical conditions like hypo- or hyperthyroidism and congenital abnormalities
12. Participation in another study with test product two months prior the study

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in stool consistency | Four weeks
  Bristol Stool Consistency Score:
  Type 1: Separate hard lumps, like nuts (hard to pass); Severe Constipation. Type 2: Sausage-shaped, but lumpy; Mild Constipation. Type 3: Like a sausage, but with cracks on its surface; Normal. Type 4: Like a sausage or snake, smooth and soft; Normal. Type 5: Soft blobs with clear-cut edges (passed easily); Borderline Normal. Type 6: Fluffy pieces with ragged edges, a mushy stool; Mild diarrhea. Type 7: Watery, no solid pieces, entirely liquid; Severe diarrhea.

SECONDARY OUTCOMES:
Change in the Frequency of Bowel Movement | four weeks
  Frequency of Bowel Movement- recorded as the number of bowel movements per day and reported as the daily average bowel movement in a week
Change in the Duration of Bowel Movement | Four weeks
  Duration of Bowel movement will be recorded in minutes in the lavatory per bowel movement per day and reported as the daily average minutes in a week.
Change in the Gastrointestinal Well-being (Patient Assessment of Constipation Symptoms) | four weeks
  This includes measures of abdominal discomfort and pain, painful bowel movement, bloating, a sense of incomplete bowel movement, straining during bowel movement, and unsuccessful bowel movement using a five-point scale (PAC-SYM).

CONTACTS AND LOCATIONS:
Overall Officials: Diane S MENDOZA-SARMIENTO, Ph.D in Health Research, Principal Investigator — University of Santo Tomas; Leslie Michelle M Dalmacio, Ph.D in Molecular Biology, Study Chair — University of the Philippines-Manila
Locations (1):
- University of Santo Tomas, Manila, Manila, Philippines

IPD SHARING:
Plan to Share IPD: No